CLINICAL TRIAL: NCT02690480
Title: Phase II Study to Compare Fulvestrant (F) 500mg Plus Placebo vs F 500mg Plus Palbociclib as First Line Treatment for Postmenopausal Women With Hormone Receptor Positive Advanced Breast Cancer Sensitive to Endocrine Therapy. GEICAM/2014-12
Brief Title: Fulvestrant (F)+Placebo vs F+Palbociclib First Line for Postmenopausal Hormone Receptor+ Advanced Breast Cancer
Acronym: FLIPPER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GEICAM/2014-12; 2015-002437-21 (EudraCT Number)
Record Dates: First submitted 2016-01-05; First posted 2016-02-24 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Breast Neoplasms
Keywords: fulvestrant; palbociclib; metastases; postmenopausal; breast cancer; hormone receptor positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — palbociclib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PD-0332991(Palbociclib)+fulvestrant(FaslodexTM) (Experimental): Fulvestrant 500mg, on days 1, 15 (±3 days) of Cycle 1, and then on Day 1 of each subsequent 28 day cycle (±3 days) in combination with Palbociclib, 125 mg, orally once daily from day 1 to day 21 followed by 7 days off treatment on every 28 days cycles.
  Interventions: Drug: PD-0332991 (Palbociclib); Drug: Fulvestrant
- Placebo+fulvestrant(FaslodexTM) (Active Comparator): Fulvestrant 500mg on days 1, 15 (±3 days) of Cycle 1, and then on Day 1 of each subsequent 28 day cycle (±3 days) in combination with Placebo orally once daily from day 1 to day 21 followed by 7 days off treatment on every 28 days cycles.
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: PD-0332991 (Palbociclib) — Palbociclib, 125 mg, orally once daily from day 1 to day 21 followed by 7 days off treatment on every 28 days cycles.
  Patients will continue to receive their assigned treatment until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first
  Other Names: Ibrance
  Arms: PD-0332991(Palbociclib)+fulvestrant(FaslodexTM)
Drug: Fulvestrant — Fulvestrant 500mg, two 5ml intramuscular injections (one in each buttock), on days 1, 15 (±3 days) of Cycle 1, and then on Day 1 of each subsequent 28 day cycle (±3 days)
  Patients will continue to receive their assigned treatment until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first
  Other Names: Faslodex
Drug: Placebo — Placebo orally once daily from day 1 to day 21 followed by 7 days off treatment on every 28 days cycles.
  Patients will continue to receive their assigned treatment until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs firs
  Arms: Placebo+fulvestrant(FaslodexTM)

SUMMARY:
This is an international, multicentre, double-blind, controlled, randomized phase II study comparing the efficacy and safety of fulvestrant in combination with palbociclib versus fulvestrant plus placebo in postmenopausal women with HR-positive/HER2-negative metastatic breast cancer who have received ≥5 years of endocrine therapy in the adjuvant setting as treatment for early disease and remained disease free for > 12 months following its completion or have "de novo" metastatic disease.

DETAILED DESCRIPTION:
Patients must have at least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline and is suitable for repeated assessment by CT, MRI or plan x-ray. Patients with bone-only disease must have a lytic or mixed (lytic + blastic) lesion, which has not been previously irradiated and can be accurately assessed by CT/MRI or x-ray. Approximately 190 patients will be randomized 1:1 between the experimental arm (approximately 95 patients treated with fulvestrant plus palbociclib) and the control arm (approximately 95 patients treated with fulvestrant plus placebo).

Primary Objective:

• To compare the efficacy of fulvestrant in combination with palbociclib versus fulvestrant plus placebo in terms of the rate of Progression-Free Survival (PFS) at 1 year in postmenopausal women with HR-positive/HER2-negative metastatic breast cancer previously treated with endocrine therapy for at least 5 years and remaining disease free for more than 12 months following its completion or have "de novo" metastatic disease

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed and dated the informed consent document and it has been obtained before conducting any procedure specifically for the study.
2. Availability of a tumor tissue sample, archival (primary tumour) or from the metastatic lesions (preferable) for the central ER, PgR and HER2 testing.
3. Histological/cytological confirmation of breast cancer with evidence of metastatic disease (loco-regional or distant), not amenable to resection or radiation therapy with curative intent.
4. Documented positive hormone receptor status (> or = 1% of tumour cells with oestrogen receptor [ER] and/or progesterone receptor [PgR] expression) based on central testing on the most recent tumour biopsy.
5. Documented HER2-negative tumour based on central testing on the most recent tumour biopsy. HER2-negative tumour is determined as immunohistochemistry score 0/1+ or negative by in situ hybridization (FISH/CISH/SISH) defined as a HER2/CEP17 ratio <2 or for single probe assessment a HER2 copy number <4.
6. Patients must have received at least 5 years of endocrine therapy in the adjuvant setting as treatment for early disease and remained disease free for more than 12 months following its completion or have "de novo" metastatic disease. Patients that have been scheduled 5 years with adjuvant endocrine therapy and stopped treatment, by patient's own decision, after completing at least 3 years of treatment, can be also be included as long as they have remained free of disease 3 years after discontinuing the endocrine therapy.
7. Patients must have at least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline and is suitable for repeated assessment by CT, MRI, plan x-ray or physical examination. Clinical lesions will only be considered measurable when they are superficial and ≥10mm diameter as assessed using callipers (e.g. skin nodules). Patients with bone-only disease must have a lytic or mixed (lytic + blastic) lesion, which has not been previously irradiated and can be accurately assessed by CT/MRI according to RECIST version 1.1.
8. Postmenopausal patient, defined as a woman fulfilling any one of the following criteria (based on the NCCN definition of menopause [National Comprehensive Cancer Network 2008]):

   * Prior bilateral oophorectomy.
   * Age > 60 years.
   * Age ≤ 60 years and with amenorrhea for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and follicle stimulating hormone and estradiol in the postmenopausal range.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2.
10. At least 18 years of age.
11. Life expectancy ≥ 12 weeks.
12. Adequate organ and bone marrow function:

    * ANC ≥ 1,500/mm3 (1.5x109/L);
    * Platelets ≥ 100,000/mm3 (100x109/L);
    * Haemoglobin (Hgb) ≥ 9g/dL (90g/L);
    * Serum creatinine ≤ 1.5xUpper Limit of Normal (ULN) or estimated creatinine clearance ≥ 60ml/min as calculated using the method standard for the institution;
    * Total serum bilirubin ≤ 1.5xULN (<3xULN if Gilbert´s disease);
    * AST and/or ALT ≤ 3xULN (≤5xULN if liver metastases present);
    * Alkaline Phosphatase (AP) ≤ 2.5xULN (≤5xULN if bone or liver metastases present).
13. Patients consent to biological sample provision for biomarker exploratory analysis.
14. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Prior systemic therapy for metastatic disease. Note: patients with a local recurrent disease treated with surgery (R0) and receiving a "second hormonal adjuvant therapy for five years" will be allowed, provided they have remained disease free for more than 12 months following its completion.
2. Have "de novo" locally advanced disease.
3. Current use of food or drugs known to be potent CYP3A4 inhibitors, drugs known to be potent CYP3A4 inducers, and drugs that are known to prolong the QT interval.
4. Presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement, or any degree of brain or leptomeningeal involvement (past or present), or symptomatic pulmonary lymphangitis spread, or any known bone marrow infiltration due to breast cancer. Patients with discrete pulmonary parenchymal metastases are eligible, provided their respiratory function is not significantly compromised as a result of disease.
5. Treatment with a non-approved or experimental drug within 4 weeks before randomization.
6. Prior treatment with any CDK4/6 inhibitor or fulvestrant.
7. Current or prior malignancy within previous 5 years (other than breast cancer or adequately treated basal cell or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix).
8. History of:

   * Bleeding diathesis (i.e., disseminated intravascular coagulation [DIC], clotting factor deficiency) or long-term (>6 months) anticoagulant therapy (other than antiplatelet therapy and low dose coumarin derivatives provided that the International Normalised Ratio (INR) is less than 1.6). Hypersensitivity to active or inactive excipients of fulvestrant, palbociclib/placebo or castor oil.
   * Any severe concomitant condition which makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the trial protocol, e.g. uncontrolled cardiac disease or uncontrolled diabetes mellitus.
9. QTc interval > 480msec, family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes.
10. Uncontrolled electrolyte disorders that can compound the effects of a QTc-prolonging drug (eg, hypocalcaemia, hypokalaemia, hypomagnesaemia).
11. Impairment of gastro-intestinal (GI) function or GI disease that may significantly alter the absorption of palbociclib, such as history of GI surgery which may result in intestinal blind loops and patients with clinically significant gastro-paresis, short bowel syndrome, unresolved nausea, vomiting, active inflammatory bowel disease or diarrhoea of CTCAE grade > 1.
12. Prior hematopoietic stem cell or bone marrow transplantation.
13. Known human immunodeficiency virus infection.
14. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of the rate of Progression-Free Survival (PFS) | at 1 year
  assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by the investigator

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | an average of 40-44 months since FPFV (approximately Ago2019)
  the time from the date of randomization to the first documented progressive disease, using RECIST version 1.1, or death from any cause, whichever occurs first
Objective Response Rate (ORR) | at 1 year and to be updated with further analyses
  the percentage of patients with a complete or partial response out of the patients who had measurable disease at baseline.
Clinical Benefit Rate (CBR) | at 1 year and to be updated with further analyses
  Complete Response (CR) plus Partial Response (PR) plus stable disease (SD) lasting ≥ 24 weeks (+/- 2 weeks) according to RECIST version 1.1.
Overall Survival (OS). | an average of 40-44 months since FPFV(approximately Ago2019). A formal analysis will be performed when at least 60% of patients have died (2021)
  the time from the date of randomization to the date of death from any cause.
1 year and 2 year survival probabilities | 1 year and 2 year
  the percentage of patients without death from any cause out of the randomised patients (calculated using the Kaplan-Meier technique).
Incidence of adverse events occurring during the study, and their relatedness to the study drug/medications (safety and tolerability). | at 1 year and to be updated with further analyses
  Safety will be assessed by standard clinical and laboratory tests. Adverse events will be graded according to NCI-CTCAE version 4.0
Patient reported outcomes of health-related quality of life based on EORTC QLQ-C30 Global Health Status/Quality of Life and Physical Function | at 1 year and to be updated with further analyses
  Generic aspects of quality of life will be assessed. Changes (mean score) from baseline and time to deterioration will be analyzed.Health Status/QoL and Physical Function and EORTC QLQ-BR23 Breast Module from baseline
Patient reported outcomes of health-related quality of life based on EORTC QLQ-BR23 Breast Module. | at 1 year and to be updated with further analyses
  Disease-specific treatment measurements will be assessed. Changes (mean score) from baseline and time to deterioration will be analyzed.

OTHER OUTCOMES:
Biomarker analyses | Up to 5 years
  Identify promising biomarkers of response to fulvestrant plus palbociclib and fulvestrant plus placebo.
  * Identify promising biomarkers of primary resistance to fulvestrant plus palbociclib and fulvestrant plus placebo.
  * Identify promising biomarkers of acquired resistance to fulvestrant plus palbociclib and fulvestrant plus placebo.
  * Identify promising biomarkers to monitor response to fulvestrant plus palbociclib and fulvestrant plus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital del Mar
Locations (32):
- Ireland (5):
  - Bon Secours Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Galway University Hospital, Galway
  - University Hospital Waterford, Waterford
- Spain (27):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Infanta Cristina, Parla, Madrid
  - Hospital Universitario Quirón de Madrid, Pozuelo de Alarcón, Madrid
  - Complejo Hospitalario Universitario Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Sant Joan Reus, Reus, Tarragona
  - Centro Oncológico de Galicia, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu y Sant Pau, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Quirón Sagrado Corazón de Sevilla, Seville
  - Hospital Universitario Vírgen del Rocío, Seville
  - Hospital Universitario de Valme, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario Valencia, Valencia
  - Hospital Universitario I Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tibau A, Martinez MT, Ramos M, De La Cruz-Merino L, Santaballa A, O'Connor M, Martinez-Janez N, Moreno F, Fernandez I, Virizuela JA, Alarcon J, de La Haba-Rodriguez J, Sanchez-Rovira P, Albacar CR, Bueno Muino C, Kelly C, Casas M, Bezares S, Rosell L, Albanell J. Quality of life with palbociclib plus fulvestrant versus placebo plus fulvestrant in postmenopausal women with endocrine-sensitive hormone receptor-positive and HER2-negative advanced breast cancer: patient-reported outcomes from the FLIPPER trial. Ther Adv Med Oncol. 2023 Jan 19;15:17588359221148921. doi: 10.1177/17588359221148921. eCollection 2023. PMID 36743520
- [Derived] Albanell J, Martinez MT, Ramos M, O'Connor M, de la Cruz-Merino L, Santaballa A, Martinez-Janez N, Moreno F, Fernandez I, Alarcon J, Virizuela JA, de la Haba-Rodriguez J, Sanchez-Rovira P, Gonzalez-Cortijo L, Margeli M, Sanchez-Munoz A, Anton A, Casas M, Bezares S, Rojo F. Randomized phase II study of fulvestrant plus palbociclib or placebo in endocrine-sensitive, hormone receptor-positive/HER2-advanced breast cancer: GEICAM/2014-12 (FLIPPER). Eur J Cancer. 2022 Jan;161:26-37. doi: 10.1016/j.ejca.2021.11.010. Epub 2021 Dec 11. PMID 34902765